CLINICAL TRIAL: NCT00781638
Title: Open Uncontrolled Investigation to Assess the Efficacy and Safety of Adacolumn® Granulocytes, Monocytes / Macrophage Apheresis Device in Children and Adolescents With Active Ulcerative Colitis
Brief Title: ADAPT Adacolumn Pediatric Trial in Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otsuka Frankfurt Research Institute GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ada-UC-08-101
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Ulcerative Colitis
Keywords: Pediatric UC, Adacolumn apheresis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Adacolumn® — The medical device Adacolumn® (CE-Mark Certificate G1 07 01 366 76013) is an adsorptive type extracorporeal apheresis column. It has been shown to effectively improve clinical and endoscopic signs and symptoms in UC in adults by removing granulocytes and monocytes and by changing the Cytokine production.
  Other Names: GMA apheresis (Granulocytes/Monocytes adsorptive apheresis).

SUMMARY:
Children aged up to 18 years with moderately active Ulcerative Colitis (PUCAI:35-64) will receive one weekly Adacolumn® apheresis treatment over 5 consecutive weeks, followed by up to 3 optional Adacolumn® apheresis treatments over 3 consecutive weeks. Primary end point is PUCAI at Week 12.

The main part of the clinical investigation will be continued by a one year follow up for responders.

DETAILED DESCRIPTION:
The individual clinical investigation period will be 12 weeks per patient. If the patient will take part in the follow up, the individual clinical investigation period will be 64 weeks.

Patients receive one weekly Adacolumn® apheresis over 5 consecutive weeks. The treating investigator may decide to add up to 3 treatments based on his judgment.

Treatment details Day -07: Screening; Day 00 Baseline: 1st Adacolumn® apheresis; Day 07: 2nd Adacolumn® apheresis; Day 14: 3rd Adacolumn® apheresis; Day 21: 4th Adacolumn® apheresis; Day 28: 5th Adacolumn® apheresis; Week 12:Final evaluation

ELIGIBILITY:
Inclusion Criteria:

1. Children and adolescents < 18 years
2. Ulcerative colitis documented by clinical symptoms, endoscopic findings and histology (in patient history)
3. Moderate active ulcerative colitis at baseline evaluation, defined as follows:PUCAI between 35 and 64
4. Pancolitis or left-sided colitis
5. Ulcerative colitis for at least 3 months
6. Receiving or having received one or more of the following medicinal products before screening:

   * Sulfasalazine, mesalamine and other 5-aminosalicylic acid (5-ASA) agents for 4 weeks or more with a stable dose for the last 2 weeks,
   * 0.5mg/kg/body weight with a maximum of 20 mg per day of prednisone with a stable dose for the last 2 weeks, or
   * 6-mercaptopurine or azathioprine for 12 weeks or more with a stable dose for the last 4 weeks Other UC medication is not allowed (see also Chapter 4.4.2).
7. For female patients of child-bearing potential, a negative pregnancy test and agreement to use an effective contraceptive method or abstain from sexual activities during the course of the clinical investigation
8. Agreement to participate in all visits
9. Signed written informed consent document by patients and their legal guardian or representative
10. Body weight must be more or equal 30kg
11. Adequate peripheral venous access to allow for completion of the apheresis treatments

Exclusion Criteria:

1. Febrile (>38ºC)
2. Evidence of toxic megacolon
3. Anticipated need for surgery within 12 weeks after Day 00
4. Major surgery within the past 6 weeks
5. Known obstructive diseases of the gastrointestinal system
6. Proctocolectomy, total colectomy, ileostomy, stoma or ileal pouch-anal anastomosis
7. A history of allergic reaction to heparin or heparin-induced thrombocytopenia
8. A history of hypersensitivity reaction associated with an apheresis procedure or intolerance of apheresis procedures
9. Known infection with enteric pathogens, pathogenic ova or parasites, or a positive assay for C. difficile toxin
10. Symptomatic hypotension
11. Pediatric heart conditions and problems at high susceptibility for thrombotic events (e.g. valve defects or similar)
12. A history of physical findings compatible with a cerebrovascular accident
13. Prosthetic heart valve, pacemaker or other permanent implant
14. Severe cardiovascular or peripheral vascular disease
15. Liver disease defined as levels of GOT [AST], GPT [ALT] or alkaline phosphatase >2.5x the upper limit of the normal range for the laboratory performing test
16. History of cirrhosis
17. Renal insufficiency, defined as serum creatinine >150% of the upper limit of the normal range for the laboratory performing the test
18. Known bleeding disorder (PT or PTT>1.5x the upper limit of the normal range for the laboratory performing the test), or concomitant anticoagulant therapy for purposes other than apheresis treatment
19. Prior history suggestive of a hypercoagulable disorder, including 1 or more episodes of pulmonary embolism or deep vein thrombosis
20. Known infection with Hepatitis B or C, or HIV
21. Abnormal hematology parameters defined as severe anemia with hemoglobin <8.5g/dL, white blood cell count of <3,500/μl and a granulocyte count <2,000/μl
22. Fibrinogen level >700mg/dL
23. Infection:

    * Active infections from successful completion of antibiotic treatment for routine bacterial infection less than 4 weeks of entry into the clinical investigation (screening)
    * Febrile viral infection within 4 weeks of entry into the clinical investigation (screening)
    * Less than 12 weeks from conclusion of therapy for systemic fungal infections to screening
24. Malignancy within the past 2 years other than surgically cured skin carcinoma or cervical dysplasia (CIN I-II)
25. History of dysplasia or carcinoma of the colon
26. Current drug or alcohol abuse
27. Pregnant, lactating or planning to become pregnant during the course of the clinical investigation
28. Used within the last 30 days an investigational medicinal product, biologic or device
29. Pre-treatment of UC with drugs other than 5-ASA and derivatives, azathioprine and or corticosteroids, e.g. immunosuppressants and biologics
30. Steroid-resistance or -dependency, defined as inability to completely withdraw steroids without inducing a relapse or flare-up of the disease
31. Topical therapy for ulcerative colitis within the last 2 weeks.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2008-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Primary response variable: Changes in mean PUCAI between baseline and Week 12 | 12 Weeks plus 1 year Follow up

SECONDARY OUTCOMES:
Difference in Endoscopic Activity Index (EAI) according to Rachmilewitz between Week 12 and baseline for those patients with 2 endoscopies | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Tarja Ruuska, MD, PhD, Principal Investigator — Tampere University Hospital